CLINICAL TRIAL: NCT04629573
Title: Epidural Anesthesia and Myomectomy-Associated Blood Loss: A Prospective Randomised Controlled Study
Brief Title: Epidural Anesthesia and Myomectomy Associated Bleeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrady S Ibrahim, MD, Professor of Anesthesia, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB0000871248
Record Dates: First submitted 2020-11-10; First posted 2020-11-16 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Epidural; Anesthesia, Headache
Keywords: Epidural anesthesia, Myomectomy
MeSH Terms: conditions — Headache | interventions — Anesthesia, General

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Epidural Anesthesia
  Interventions: Procedure: Lumber Epidural
- Group 2 (Active Comparator): General Anesthesia
  Interventions: Procedure: General anesthesia

INTERVENTIONS:
Procedure: Lumber Epidural — Epidural procedure was performed by attending anesthesiologists who had completed at least 50 epidural procedures during their training. Patient was placed in the sitting position, the skin over the lumbar area was cleaned and a sterile technique was observed throughout the procedure. Skin and subcutaneous tissue were infiltrated with 1% lidocaine 2 mL at the intended site of epidural placement (L2-3 or L3-4 interspace). The lumbar epidural space was then located, using a midline approach with an 18 gauge Tuohy epidural needle via a loss of resistance technique with 2 mL of saline, 20 gauge epidural catheter was placed in each patient. We deliver an initial bolus of 20 ml bupivacaine 0.5% plus 100 mcg Fentanyl, followed by continuous infusion of bupivacaine 0.5% plus 1mcg/ml Fentanyl (3-5 ml/hr.).
  Arms: Group 1
Procedure: General anesthesia — Anesthesia was initiated with IV fentanyl 1 µg/kg, propofol 2 mg/kg and cisatracurium 0.15 mg/kg to facilitate endotracheal intubation. After tracheal intubation, anesthesia was maintained with sevoflurane in O2 and air (FiO2 of 0.5), cisatracurium 1µg/kg/min and fentanyl 0.5 µg/ kg /h were infused. Volume-Controlled ventilation was performed in all patients. Cisatracurium and fentanyl infusion was stopped at the end of surgery, neuromuscular blockade was reversed, and the patient was extubated and send to post-anesthesia care unit.
  Arms: Group 2

SUMMARY:
This is a prospective study for abdominal myomectomies performed from June 2012 to June 2019 by a single surgeon in a tertiary care referral hospital. Large uterine myoma was defined as the estimated diameter of dominant myoma equal to or larger than 10 cm by sonography. Demographics, diagnosis, perioperative variables, operative outcomes and complications were recorded. The Intraoperative anesthetic management, blood and blood products transfusion, and total volume of blood loss, as well as postoperative follow-up, were reviewed for each patient.

DETAILED DESCRIPTION:
Randomization and Blinding: To allow randomization, researchers prepared the management protocol for each group and sealed one protocol per envelope with a computer-generated number assigned prior to study initiation. Randomization was performed by picking the numbered study envelopes sequentially and opened before induction of anesthesia by the anesthesia doctor and managing the participant based on the enclosed protocol. The study will not be double-blinded, as it is impossible to blind the health care workers and women involved for the strategy to which the woman is allocated.

Interventions Anesthesia technique: On arrival to the operative theatre, an 18 gauge IV catheter was inserted and 500 ml of NaCl (0.9%) was infused, 1 mg midazolam was administered iv as premedication. Patients were monitored with continuous electrocardiography and pulse oximetry and intermittent non-invasive blood pressure measurements every 5 min.

Lumbar epidural: Epidural procedure was performed by attending anesthesiologists who had completed at least 50 epidural procedures during their training. Patient was placed in the sitting position, the skin over the lumbar area was cleaned and a sterile technique was observed throughout the procedure. Skin and subcutaneous tissue were infiltrated with 1% lidocaine 2 mL at the intended site of epidural placement (L2-3 or L3-4 interspace). The lumbar epidural space was then located, using a midline approach with an 18 gauge Tuohy epidural needle via a loss of resistance technique with 2 mL of saline, 20 gauge epidural catheter was placed in each patient. We deliver an initial bolus of 20 ml bupivacaine 0.5% plus 100 mcg Fentanyl, followed by continuous infusion of bupivacaine 0.5% plus 1mcg/ml Fentanyl (3-5 ml/hr.).

General anesthesia: Anesthesia was initiated with IV fentanyl 1 µg/kg, propofol 2 mg/kg and cisatracurium 0.15 mg/kg to facilitate endotracheal intubation. After tracheal intubation, anesthesia was maintained with sevoflurane in O2 and air (FiO2 of 0.5), cisatracurium 1µg/kg/min and fentanyl 0.5 µg/ kg /h were infused. Volume-Controlled ventilation was performed in all patients. Cisatracurium and fentanyl infusion was stopped at the end of surgery, neuromuscular blockade was reversed, and the patient was extubated and send to post-anesthesia care unit.

Myomectomy: Abdominal myomectomy was performed in the standard conventional fashion. A single surgeon handled all the surgical procedures. The myomectomy was performed by enucleating the fibroid and closing the uterine defect in multiple layers. The use of energy devices, suture type, and adhesion barriers were at the discretion of the surgeon.

ELIGIBILITY:
Inclusion Criteria

* Women over 18 years old
* American Society of Anesthesiologist (ASA) I and II
* Undergoing myomectomy for treatment of large uterine leiomyomas with a minimum diameter of 10 cm

Exclusion Criteria:

* Patients with previous uterine surgery (myomectomy, cesarean delivery)
* Coagulopathy or other bleeding diathesis
* Severe anemia (Hb under 5.0 g/dl)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 78 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Blood loss | 24 hours
  Intraoperative blood loss

CONTACTS AND LOCATIONS:
Overall Officials: Abdelrady S Ibrahim, Principal Investigator — Assiut University
Locations (1):
- Assiut university faculty of medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhang Y, Yu J, Yang F, Zhao L, Ma L, Zhang H, Chen X, Ma H. Effect of anesthetic technique on serum vascular endothelial growth factor C and prostaglandin E2 levels in women undergoing surgery for uterine leiomyomas. J Int Med Res. 2020 Apr;48(4):300060520918420. doi: 10.1177/0300060520918420. PMID 32314939